CLINICAL TRIAL: NCT00947206
Title: Lay Health Workers and Colorectal Cancer Screening Among Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco State University (Other); NICOS Chinese Health Coalition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA138778-01A1 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Neoplasms
Keywords: Chinese Americans; lay health worker outreach; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LHWO about CRC (Experimental): The intervention group participants will be exposed to 2 LHWO sessions and 2 telephone calls aimed at increasing their CRC screening receipt.
  Interventions: Behavioral: LHWO about CRC
- Nutrition education + CRC brochure (Active Comparator): The comparison group will receive a bilingual CRC brochure as well as a lecture on healthy nutrition for cardiovascular health and a post-intervention LHWO session on CRC screening.
  Interventions: Behavioral: Nutrition Education + CRC brochure

INTERVENTIONS:
Behavioral: LHWO about CRC — 2 LHWO sessions and 2 telephone calls aimed at increasing their CRC screening receipt
  Arms: LHWO about CRC
Behavioral: Nutrition Education + CRC brochure — Bilingual CRC brochure as well as a lecture on healthy nutrition for cardiovascular health and a post-intervention LHWO session on CRC screening.
  Arms: Nutrition education + CRC brochure

SUMMARY:
This proposed project seeks to expand understanding of what constitutes a "lay health worker (LHW)," how those characteristics determine the effectiveness of LHWs as health educators on colorectal cancer (CRC) screening, and the relationship of those characteristics to a particular community and culture. Using quantitative and qualitative methods and a community-based participatory research (CBPR) approach, the project will develop and implement a group randomized controlled trial to evaluate LHW effectiveness in promoting CRC screening among Chinese Americans age 50 to 75 with a pilot component to evaluate the role of Traditional Chinese Medicine (TCM) healers as health educators.

The investigators will conduct focus groups with community participants to revise training materials developed in a prior pilot project. The investigators will also conduct ethnographic observations of TCM healers and focus groups with their clients to refine the training materials. The investigators will recruit 26 LHWs to be assigned to the intervention arm and 26 to the comparison arm. The LHWs will each recruit 12 participants from their social network for a total of 312 participants in each arm. The intervention group participants will be exposed to 2 LHWO sessions and 2 telephone calls aimed at increasing their CRC screening receipt. The comparison group will receive a bilingual CRC brochure as well as a lecture on healthy nutrition for cardiovascular health and a post-intervention LHWO session on CRC screening. Effectiveness of the intervention will be measured by pre-intervention and post-intervention surveys of community participants' CRC screening behaviors, with validation of self-reports. An additional 10 TCM healers will also participate as LHWs. They will each recruit 12 participants for LHWO. There will be extensive ethnographic observations as well as post-intervention focus groups of LHWO activities, LHWs, and LHWO participants to assess the factors that contribute to effective LHWO.

The primary hypothesis is that the increase in the proportion of participants who report ever having had a CRC screening test in the experimental group (LHWO about CRC) will be greater than the increase in the comparison group (nutrition education + CRC brochure).

DETAILED DESCRIPTION:
The secondary hypotheses are:

1. The increase in the proportion of participants who are up-to-date for CRC screening in the experimental group will be greater than the increase in the comparison group;
2. The increase in the proportion of participants who intend to obtain CRC screening in the next 6 months in the experimental group will be greater than the increase in the comparison group;
3. The increase in the proportion of participants who are aware of CRC screening tests in the experimental group will be greater than the increase in the comparison group;
4. Self-efficacy is a mediator between intervention and receipt of CRC screening.
5. Knowledge is a mediator between intervention and receipt of CRC screening.
6. Gender is a moderator between intervention and receipt of CRC screening.

Although the pilot project intervention was effective in both men and women, the sample was too small to determine if there was a gender effect. Based on the extensive literature on LHWO among women, the intervention may be more effective among women than men.

Additional secondary hypotheses will apply the primary hypothesis and secondary hypotheses 1-3 to individual CRC tests (FOBT, sigmoidoscopy, or colonoscopy) rather than to the combined outcome.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Chinese or Chinese Americans
* age 50 to 75
* speak a language that the LHW can speak (Cantonese, Mandarin, and/or English)
* live and intend to stay in SF for at least 12 months
* have no personal history of CRC
* have no medical problems preventing them from attending educational sessions
* willing to participate in a study about health behaviors involving nutrition or CRC screening

Exclusion Criteria:

* anyone who does not meet the above criteria
* those unable to understand informed consent form written in their language
* those too debilitated to attend educational sessions

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 909 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
ever had a CRC screening test | 6 months

SECONDARY OUTCOMES:
up-to-date for CRC screening | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tung T Nguyen, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - NICOS, San Francisco, California
  - San Francisco State University, San Francisco, California

REFERENCES:
- [Background] Wong ST, Gildengorin G, Nguyen T, Mock J. Disparities in colorectal cancer screening rates among Asian Americans and non-Latino whites. Cancer. 2005 Dec 15;104(12 Suppl):2940-7. doi: 10.1002/cncr.21521. PMID 16276538
- [Background] Mock J, McPhee SJ, Nguyen T, Wong C, Doan H, Lai KQ, Nguyen KH, Nguyen TT, Bui-Tong N. Effective lay health worker outreach and media-based education for promoting cervical cancer screening among Vietnamese American women. Am J Public Health. 2007 Sep;97(9):1693-700. doi: 10.2105/AJPH.2006.086470. Epub 2007 Feb 28. PMID 17329652
- [Background] Wu AP, Burke A, LeBaron S. Use of traditional medicine by immigrant Chinese patients. Fam Med. 2007 Mar;39(3):195-200. PMID 17323211
- [Background] Nguyen TT, Love MB, Liang C, Fung LC, Nguyen T, Wong C, Gildengorin G, Woo K. A pilot study of lay health worker outreach and colorectal cancer screening among Chinese Americans. J Cancer Educ. 2010 Sep;25(3):405-12. doi: 10.1007/s13187-010-0064-3. Epub 2010 Mar 5. PMID 20204570
- [Derived] Nguyen TT, Tsoh JY, Woo K, Stewart SL, Le GM, Burke A, Gildengorin G, Pasick RJ, Wang J, Chan E, Fung LC, Jih J, McPhee SJ. Colorectal Cancer Screening and Chinese Americans: Efficacy of Lay Health Worker Outreach and Print Materials. Am J Prev Med. 2017 Mar;52(3):e67-e76. doi: 10.1016/j.amepre.2016.10.003. Epub 2016 Dec 13. PMID 27986352